CLINICAL TRIAL: NCT00478322
Title: Pharmacodynamic Study of the Effect of INCB013739 on Insulin Sensitivity in Obese, Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 13739-201
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Diabetes;; Type II diabetes;; Non-insulin dependent diabetes;; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- INCB013739 (Experimental)
  Interventions: Drug: INCB013739
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo of 100 mg BID
  Arms: Matching Placebo
Drug: INCB013739 — INCB013739 100 mg BID
  Arms: INCB013739

SUMMARY:
Purpose: A 28-day US study in patients with type 2 diabetes mellitus to assess the safety and tolerability as well as the effects of treatment with an investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Have an established diagnosis of Type 2 Diabetes as determined by the investigator.
2. Females will be postmenopausal for at least 1 year with documented FSH > 30 IU/L.

Exclusion Criteria:

1. Hypertriglyceridemia > 500 mg/dL at screening.
2. BMI > 40 kg/m2.
3. Receiving thiazolidinediones, insulin, or exenatide within the 3 months prior to screening.
4. History or clinical manifestations of Addison's disease, Cushing's Syndrome, or other disorders involving glucocorticoids or mineralocorticoids.
5. Current treatment or treatment within 30 days or five half-lives (whichever is longer) prior to the first dose of study medication with another investigational medication or current enrollment in another investigational protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Changes in lipid profile laboratory values | Measured at baseline and weekly for four weeks
Assessment of pharmacokinetics of INCB013739 through analysis of blood samples. | Measured at baseline and weekly for four weeks
Assessment of pharmacodynamics of INCB013739 through analysis of blood samples | Measured at baseline and weekly for four weeks
Assessment of ECGs, physical examinations and laboratory values for adverse events | Measured at baseline through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Study Director — Incyte Corporation
Locations (3):
- United States (3):
  - Chula Vista, California
  - The Bronx, New York
  - San Antonio, Texas